CLINICAL TRIAL: NCT04415554
Title: The Effect of Aminoglycosides on Ductus in Preterm Infants
Brief Title: Aminoglycosides and Duct
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Ayala Gover, Neonatologist, Carmel Medical Center
Other Study IDs: CMC-19-0110-CTIL
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Patent Ductus Arteriosus
MeSH Terms: conditions — Ductus Arteriosus, Patent | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- exposure to aminoglicosides: preterm receiving aminoglycosides
  Interventions: Diagnostic Test: echocardiography
- non exposure to aminoglycosides: preterm not receiving aminoglycosides
  Interventions: Diagnostic Test: echocardiography

INTERVENTIONS:
Diagnostic Test: echocardiography — echocardiography exam of the infant

SUMMARY:
The aim of the study is to assess the effect of aminoglycoside treatment on ductal closure in preterms

ELIGIBILITY:
Inclusion Criteria:

infants born at or above 32 weeks of gestation

-

Exclusion Criteria:

* infants who are unlikely to survive or have congenital heart defects

Ages: 30 Minutes to 3 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: preterm infants hospitalized in NICU
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
ductal closure | 3 weeks
  closure of ductus arteriosus